CLINICAL TRIAL: NCT06179199
Title: Evaluation of the Analgesic Effect of Transcranial Direct Current Stimulation (tDCS) for Sedated Patients in Intensive Care Unit.Randomized, Placebo-controlled, Double-blind Study.
Brief Title: Evaluation of the Analgesic Effect of Transcranial Direct Current Stimulation (tDCS) for Sedated Patients in Intensive Care Unit.
Acronym: REASTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 38RC23.0217
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Transcranial Direct Current Stimulation (tDCS)
Keywords: Pain management; Transcranial direct current stimulation (tDCS); Analgesic therapy; Chronic pain; Sedated patient; Intensive care unit
MeSH Terms: conditions — Agnosia; Chronic Pain

STUDY DESIGN:
Intervention Model Description: * Active tDCS stimulation ;
  * Placebo tDCS stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS stimulation (Experimental)
  Interventions: Device: SOOMA™ tDCS™
- Placebo tDCS stimulation (Placebo Comparator)
  Interventions: Device: SOOMA™ tDCS™

INTERVENTIONS:
Device: SOOMA™ tDCS™ — The SOOMA™ tDCS™ device is designed to treat chronic pain, with a stimulation current of 2milliampere and a duration of 20 minutes

SUMMARY:
Pain management for sedated ICU patients is complex, partly because of the difficulty of assessing pain in non-communicative patients, and partly because of the side effects associated with excessive use of morphine.

In this context, the use of another non-pharmacological approach, transcranial direct current stimulation (tDCS), could be of interest. With tDCS, neuronal activity is modulated by inducing a weak electric current through the cerebral cortex between two electrodes applied to the surface of the scalp. Although the mechanisms of action of tDCS are not yet fully understood, the medium-term effects are thought to be linked to the activation of N-methyl-D-aspartate receptors, glutamate-activated receptors involved in cellular memory. The use of tDCS as an analgesic therapy for chronic pain has produced encouraging results in patients suffering from fibromyalgia, migraine and central pain following spinal cord injury, Its use in sedated intensive care patients is unknown. To assess the possible analgesic effect of tDCS in these patients, we will use quantitative pupillometry, a technique already used in routine intensive care, to quantify nociception during a standardized nociceptive simulation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 80 years,
* Sedated patient requiring mechanical ventilation for at least 48 hours with administration of morphine.
* Person affiliated to the social security system or beneficiary of an assimilated regime.
* RASS ≤ -2
* Close consent or emergency inclusion

Exclusion Criteria:

* History of epilepsy.
* Severe brain injury (head trauma, stroke, neuromeningeal infection, status epilepticus).
* Presence of intracranial ferromagnetic material.
* Presence of electronic stimulators or implants (e.g. pacemaker, spinal cord or intracranial stimulator).
* Facial trauma preventing eye opening.
* Patients who are blind and/or have eye damage.
* Protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons under legal protection.
* Subjects excluded from another study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pupillary Pain Index measurement | From Day1 to Day 4
  Measurement of the Pupillary Pain Index before and at the end of the tDCS stimulation session in both groups (active stimulation or placebo)

SECONDARY OUTCOMES:
Comparison between groups of daily consumption of analgesics and sedatives | From Day1 to Day 4
Inter-group comparison of changes in Behavioral Pain Scale score during painful care (tracheal suctioning) | From Day1 to Day 4
Inter-group comparison of variations in pupil diameter measured by quantitative pupillometry in response to painful care (tracheal suctioning). | From Day1 to Day 4
Inter-group comparison of changes in sedation levels measured by the Richmond Agitation-Sedation Scale | From Day1 to Day 4
Inter-group comparison of the proportion of patients with a reduction in the Pupillary Pain Index ≥2 from baseline at the end of treatment. | From Day1 to Day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Management Center - Chuga, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Pinto CB, Teixeira Costa B, Duarte D, Fregni F. Transcranial Direct Current Stimulation as a Therapeutic Tool for Chronic Pain. J ECT. 2018 Sep;34(3):e36-e50. doi: 10.1097/YCT.0000000000000518. PMID 29952860
- [Background] Payen JF, Bru O, Bosson JL, Lagrasta A, Novel E, Deschaux I, Lavagne P, Jacquot C. Assessing pain in critically ill sedated patients by using a behavioral pain scale. Crit Care Med. 2001 Dec;29(12):2258-63. doi: 10.1097/00003246-200112000-00004. PMID 11801819